CLINICAL TRIAL: NCT05295498
Title: Analgesic Effect of Accelerated Repetitive Transcranial Magnetic Stimulation in Pain Related to Peripheral Neuropathy
Brief Title: Analgesic Effect of Accelerated Repetitive Transcranial Magnetic Stimulation in Neuropathic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jakub Antczak (Other)
Responsible Party: Sponsor-Investigator, Jakub Antczak, Principal Investigator, Jagiellonian University
Organization: Jagiellonian University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JagiellonianU69
Record Dates: First submitted 2022-03-07; First posted 2022-03-25 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Neuropathy
Keywords: Peripheral neuropathy; Neuropathic pain; rTMS; analgesic effect
MeSH Terms: conditions — Peripheral Nervous System Diseases; Neuralgia

STUDY DESIGN:
Intervention Model Description: Parallel Assignment. Patients will be randomly assigned to active or to sham stimulation.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcomes Assessor). Sham stimulation will be provided by holding the stimulating coil perpendicularly to the scalp, which assures similar impression as during active stimulation but prevents significant magnetic field to reach the brain tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active repetitive transcranial magnetic stimulation (Experimental): 10 hertz (Hz) rTMS will be administered over the primary motor area. Therapy will include 6 sessions (three sessions in two consecutive days). In every sessions 1500 magnetic pulses of 90% of the resting motor threshold intensity will be elicited.
  Interventions: Device: Active repetitive transcranial magnetic stimulation
- Sham repetitive transcranial magnetic stimulation (Sham Comparator): Sham stimulation will mimic the active one except that the stimulating coil will be held perpendicularly to the scalp, which assures similar impression as the active stimulation but prevents that significant magnetic field will reach brain tissue.
  Interventions: Device: Sham repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Active repetitive transcranial magnetic stimulation — High frequency rTMS over the primary motor area to induce the long term potentiation of primary motor areas for the muscles of upper extremity.
  Arms: Active repetitive transcranial magnetic stimulation
Device: Sham repetitive transcranial magnetic stimulation — Sham stimulation to mimic the high frequency rTMS over the primary motor area.
  Arms: Sham repetitive transcranial magnetic stimulation

SUMMARY:
Peripheral neuropathy is a frequent condition, commonly associated with pain. Repetitive Transcranial Magnetic Stimulation (rTMS) is a noninvasive method of modulation of brain plasticity and is regarded as one of alternative methods to alleviate pain associated with various kind of neuropathies. rTMS is usually performed once a day and the whole therapy of neuropathic pain lasts one week. In a number of recent clinical trials including patients with depression and some other disorders, rTMS was delivered several times a day, which reduced the time of the whole therapy. This approach was termed an accelerated rTMS. The purpose of this study is to investigate feasibility of accelerated rTMS in treatment of neuropathic pain.

DETAILED DESCRIPTION:
Peripheral neuropathy is a frequent condition, commonly associated with pain, which is often drug resistant. Repetitive Transcranial Magnetic Stimulation (rTMS) is a noninvasive method of modulation of brain plasticity. In this method, series of magnetic stimuli are delivered to the cerebral cortex, where they turn to electric current and depolarize repetitively the targeted neurons. If the stimulation is repeated during subsequent days it is capable to modify the activity of targeted cortical area for weeks or even months and by this way to achieve therapeutic effect. rTMS is most commonly used to treat drug-resistant depression but a number of other psychiatric and neurologic conditions is increasingly being regarded as therapeutic indication for rTMS. In patients suffering from neuropathic pain rTMS is delivered with high frequency, over primary motor areas (PMA). Stimulation of PMA should result in modulation of thalamic activity, achieved by antidromic excitation of thalamocortical connections. rTMS is usually performed once a day and the whole therapy of neuropathic pain lasts one week. In a number of recent clinical trials including patients with depression and some other disorders, rTMS was delivered several times a day, which reduced the time of the whole therapy. This approach was termed an accelerated rTMS. The purpose of this study is to investigate feasibility of accelerated rTMS in treatment of neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of peripheral neuropathy
* Neuropathic pain of constant severity since not less than a month and requiring use of analgesics more than once a week
* Score of 30 millimeter or more on the 100 millimeter visual analog scale of pain intensity at inclusion

Exclusion Criteria:

* Severe depression
* Personality disorders and other psychiatric conditions, which could disturb the participation in the study
* Cognitive deficits, which could disturb the participation in the study
* Epilepsy
* Presence of magnetic material in the reach of magnetic field
* Pregnancy
* Likelihood to get pregnant
* Intracranial electrodes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale of Pain Severity after rTMS | Through study completion, an average of 1 year.
  An analog scale of the length of 100 millimeter. Total score of 100, with higher scores representing more severe pain. Change from baseline score in the Visual Analogue Scale to the measurement taken after finishing rTMS.
Visual Analogue Scale of Pain Severity First Follow-up | Before rTMS, up to one day after finishing rTMS.
  An analog scale of the length of 100 millimeter. Total score of 100, with higher scores representing more severe pain. Change from baseline score in the Visual Analogue Scale to the measurement taken after two weeks after finishing rTMS.
Visual Analogue Scale of Pain Severity Second Follow-up | Before rTMS, four weeks after finishing rTMS.
  An analog scale of the length of 100 millimeter. Total score of 100, with higher scores representing more severe pain. Change from baseline score in the Visual Analogue Scale to the measurement taken after four weeks after finishing rTMS.

SECONDARY OUTCOMES:
Numeric Pain Severity Scale after rTMS | Before rTMS, up to one day after finishing rTMS.
  Total score 10, with higher scores representing more severe pain. Change from baseline score in the Numeric Pain Severity Scale to the measurement taken after finishing rTMS.
Numeric Pain Severity Scale First Follow-up | Before rTMS, two weeks after finishing rTMS.
  Total score 10, with higher scores representing more severe pain. Change from baseline score in the Numeric Pain Severity Scale to the measurement taken two weeks after finishing rTMS.
Numeric Pain Severity Scale Second Follow-up | Before rTMS, four weeks after finishing rTMS.
  Total score 10, with higher scores representing more severe pain. Change from baseline score in the Numeric Pain Severity Scale to the measurement taken after four weeks after finishing rTMS.
Neuropathic Pain Symptoms Inventory after rTMS | Before rTMS, up to one day after finishing rTMS.
  Total score 120, with higher scores representing more severe pain and other symptoms of neuropathy. Change from baseline score in the Neuropathic Pain Symptoms Inventory to the measurement taken after finishing rTMS.
Neuropathic Pain Symptoms Inventory First Follow-up | Before rTMS, two weeks after finishing rTMS.
  Total score 120, with higher scores representing more severe pain and other symptoms of neuropathy. Change from baseline score in the Neuropathic Pain Symptoms Inventory to the measurement taken two weeks after finishing rTMS.
Neuropathic Pain Symptoms Inventory Second Follow-up | Before rTMS, four weeks after finishing rTMS.
  Total score 120, with higher scores representing more severe pain and other symptoms of neuropathy. Change from baseline score in the Neuropathic Pain Symptoms Inventory to the measurement taken four weeks after finishing rTMS.
Athens Insomnia Scale after rTMS | Before rTMS, up to one day after finishing rTMS.
  Total score 24, with higher scores representing more severe insomnia. Change from baseline score in the Athens Insomnia Scale to the measurement taken after finishing rTMS.
Athens Insomnia Scale First Follow-up | Before rTMS, two weeks after finishing rTMS.
  Total score 24, with higher scores representing more severe insomnia. Change from baseline score in the Athens Insomnia Scale to the measurement taken two weeks after finishing rTMS.
Athens Insomnia Scale Second Follow-up | Before rTMS, four weeks after finishing rTMS.
  Total score 24, with higher scores representing more severe insomnia. Change from baseline score in the Athens Insomnia Scale to the measurement taken four weeks after finishing rTMS.
Bilateral Dynamometric Assessment of the strength of the foot extension after rTMS | Before rTMS, up to one day after finishing rTMS.
  Change from baseline strength of the foot extension to the measurement taken after finishing rTMS.
Bilateral Dynamometric Assessment of the strength of the foot extension First Follow-up | Before rTMS, two weeks after finishing rTMS.
  Change from baseline strength of the foot extension to the measurement taken two weeks after finishing rTMS.
Bilateral Dynamometric Assessment of the strength of the foot extension Second Follow-up | Before rTMS, four weeks after finishing rTMS.
  Change from baseline strength of the foot extension to the measurement taken four weeks after finishing rTMS.

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Klupa, Professor, Study Chair — Jagiellonian University
Locations (1):
- Jagiellonian University Medical College, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Yes
After completing the study, the age and gender of participants as well as the scores and results of all outcome measurements made at baseline, after rTMS, at the first and at the second follow-up will be made available to other researchers on request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available after the study results will be published.
Access Criteria: On request sent by e-mail to jakub.antczak@uj.edu.pl